CLINICAL TRIAL: NCT06730061
Title: A Phase III, Open-label, Single Arm Study to Investigate the Efficacy and Safety of Elafibranor 80 mg in Adult Japanese Participants With Primary Biliary Cholangitis (PBC)
Brief Title: A Study of Elafibranor in Adult Japanese Participants With Primary Biliary Cholangitis (PBC)
Acronym: ELONSEN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-60190-462
Record Dates: First submitted 2024-12-03; First posted 2024-12-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elafibranor (Experimental): Participants will take the study intervention by mouth (swallow whole) once daily
  Interventions: Drug: Elafibranor

INTERVENTIONS:
Drug: Elafibranor — Tablet of 80 mg

SUMMARY:
The purpose of this study is to find out about the safety and how well the study intervention (elafibranor) works in participants with PBC. The participants in this study will have confirmed PBC with inadequate response or intolerance to UDCA, which is a medication used in the management and treatment of cholestatic liver disease.

PBC is a slowly progressive disease characterised by damage of the bile ducts in the liver, leading to a build-up of bile acids which causes further damage. The liver damage in PBC may lead to scarring (cirrhosis).

PBC may also be associated with multiple symptoms. Many patients with PBC may require a liver transplant or may die if the disease progresses and a liver transplant is not done. In this study all participants will receive a daily dose of elafibranor (the study intervention).

The main aim of this study is to determine if elafibranor reduces alkaline phosphatase (ALP) and total bilirubin levels. High ALP and bilirubin levels in the blood can indicate liver disease.

There will be 4 periods in this study: A screening period (up to 10 weeks) to assess whether the participant can take part. A treatment period (52 weeks) where all eligible participants will receive elafibranor. A variable treatment extension period (2-5 years) from End Of Treatment (EOT) period up to the commercial availability of elafibranor in Japan. A follow-up period (4 weeks) where participants' health will be monitored.

Participants will undergo blood sampling, urine collections, physical examinations, clinical evaluations, electrocardiograms (ECG: recording of the electrical activity of heart), ultrasound examinations (a non-invasive test that passes a probe over skin to look at the bladder, urinary tract, and liver), and Fibroscan® examinations (to measure stiffness of the liver). They will also be asked to fill in questionnaires. Each participant will be in this study for up to approximately 6 years

ELIGIBILITY:
Inclusion Criteria:

* Must have provided written informed consent and agree to comply with the study protocol.
* Japanese male or female participants aged 18 to 75 years inclusive at Screening Visit 1 (SV1).
* PBC diagnosis as described in the study protocol
* ALP ≥1.67×ULN (mean value based on samples collected at SV1 and SV2).
* TB ≤2×ULN at SV1 and SV2.
* Must have at least 4 available values for PBC Worst Itch Numeric Rating Scale (NRS) during each of the 7-day intervals in the 14 days prior to visit (V)1, for a total of at least 8 values for PBC Worst Itch NRS in the last 14 days prior to V1.
* Participants taking UDCA for at least 12 months (stable dose ≥3 months) prior to screening, or unable to tolerate UDCA treatment (no UDCA for ≥3 months) prior to screening (per country standard-of-care dosing).
* If on colchicine, must be on a stable dose for ≥3 months prior to screening.
* Medications for management of pruritus (for example, cholestyramine, rifampicin, naltrexone, sertraline or nalfurafine hydrochloride) must be on a stable dose for ≥3 months prior to screening.
* Participants taking statins or ezetimibe must be on a stable dose for ≥2 months prior to screening.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

Exclusion Criteria

* History or presence of other concomitant liver disease
* Participants with known cirrhosis who have a Child-Pugh B or C classification.
* Participants with cirrhosis with Child-Pugh A classification are allowed.
* History or presence of clinically significant hepatic decompensation,
* Medical conditions that may cause non-hepatic increases in ALP (for example, Paget's disease) or which may diminish life expectancy to <2 years, including known cancers.
* Known malignancy or history of malignancy within the last 5 years, with the exception of local, successfully treated basal cell carcinoma or in-situ carcinoma of the uterine cervix.
* Participant has a positive test for human immunodeficiency virus (HIV) Type 1 or 2 at screening, or participant is known to have tested positive for HIV.
* Evidence of any other unstable or untreated clinically significant immunological, endocrine, haematologic, gastrointestinal, neurological, or psychiatric disease as evaluated by the investigator; other clinically significant medical conditions that are not well controlled.
* History of alcohol abuse, defined as consumption of more than 30 g pure alcohol per day for men, and more than 20 g pure alcohol per day for women, or other substance abuse within 1 year prior to SV1.
* For female participants: known pregnancy, or has a positive serum pregnancy test, or breastfeeding.
* Administration of the following medications are prohibited as specified below:

  1. 1 month prior to screening: fibrates.
  2. 2 months prior to screening: glitazones.
  3. For participants with previous exposure to obeticholic acid (OCA), OCA should be discontinued 3 months prior to screening.
  4. 3 months prior to screening: azathioprine, cyclosporine (systemic), methotrexate, mycophenolate, pentoxifylline, budesonide and other systemic corticosteroids (parenteral and oral chronic administration only); potentially hepatotoxic drugs (including α-methyldopa, sodium valproate/valproic acid isoniazid, or nitrofurantoin).
  5. 12 months prior to screening: antibodies or immunotherapy directed against interleukins (ILs) or other cytokines or chemokines.
* Participants who are currently participating in, plan to participate in, or have participated in an investigational drug study or medical device study containing active substance within 30 days or 5 half-lives, whichever is longer, prior to screening; for participants with previous exposure to seladelpar, seladelpar should be discontinued 3 months prior to screening.
* Participants with previous exposure to elafibranor.
* SV1 or SV2 value ALT and/or AST >5×ULN.
* For participants with aminotransferases or TB >ULN at SV1, variability (between SV1 and SV2) of aminotransferases or TB >40%.
* SV1 value albumin <3.0 g/dL.
* Severely advanced participants according to Rotterdam criteria (TB >ULN and albumin <LLN).
* SV1 international normalised ratio (INR) >1.3 due to altered hepatic function.
* SV1 creatine phosphokinase (CPK) >2×ULN.
* SV1 serum creatinine >1.5 mg/dL.
* Significant renal disease, including nephritic syndrome, chronic kidney disease (defined as participants with markers of kidney failure damage or estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2) calculated by modification of diet in renal disease study (MDRD).
* SV1 platelet count <150×103/μL.
* Alpha-fetoprotein (AFP) >20 ng/mL with 4-phase liver computerised tomography (CT) or magnetic resonance imaging (MRI) imaging suggesting presence of liver cancer.
* Known hypersensitivity to the investigational product or to any of the formulation excipients of the elafibranor tablet.
* Mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-12-17 (Estimated); Study Completion 2032-04-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with Alkaline phosphatase (ALP) <1.67x ULN, ALP decrease ≥15% and Total Bilirubin (TB) ≤ ULN | At Week 52

SECONDARY OUTCOMES:
Percentage of Participants who normalised ALP Levels | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Change from baseline in ALP Levels | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Percentage of Participants With ALP Level response | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  Defined as 10%, 20% and 40% ALP reduction from baseline
Percentage of participants with ALP <1.5×ULN, ALP decrease ≥40% and TB ≤ULN. | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Percentage of participants with ALP <3×ULN, aspartate aminotransferase (AST) <2×ULN and Total Bilirubin (TB) <1 mg/dL (Paris I criteria). | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Percentage of participants with ALP ≤1.5×ULN, AST ≤1.5×ULN and TB ≤ULN (Paris II criteria). | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Percentage of participants with TB response rate of 15% change. | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Percentage of participants with normalisation of abnormal TB and/or albumin (Rotterdam criteria). | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Percentage of participants with TB ≤0.6×ULN | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Percentage of participants with ALP ≤1.67×ULN and TB ≤1 mg/dL. | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Percentage of participants with no worsening of TB Levels | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Percentage of participants with complete biochemical response | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  Defined as normal ALP; TB; AST; alanine aminotransferase (ALT); albumin; and INR.
Percentage of participants with ALP ≤1.67×ULN, ALP decrease ≥15% and TB ≤ULN. | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Percentage of participants with ALP <1.5×ULN, ALP decrease ≥15% and TB ≤ULN. | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Percentage of participants with ALP ≤ULN and TB ≤ULN. | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Change from baseline in PBC risk scores based in Global PBC Study Group (GLOBE) score | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  The GLOBE score is a validated risk assessment tool providing an estimate of transplant-free survival for patients with PBC. It was developed by the Global PBC Study Group using Cox regression model on over 4,000 patients with PBC. Lower GLOBE score predicts lower risk.
Change from baseline in PBC risk scores based on United Kingdom (UK)-PBC score. | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  PBC risk score developed by United Kingdom (UK)-PBC Consortium is a scoring system and the calculation is based on laboratory test measurements and upper limits of normal (ULN) for the total bilirubin (BIL12); alanine transaminase or aspartate transaminase (TA12), and alkaline phosphatase (ALP12) after at least 12 months of UDCA, and the laboratory test measurements and lower limits of normal (LLN) for the serum albumin and platelet count in the same timeframe. A high number is indicative of a worse score.
Response based on the normalisation of bilirubin. | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Response based on the normalisation of albumin Levels. | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Change from baseline in hepatobiliary injury and liver function | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  Hepatobiliary injury and liver function will be measured by AST, ALT, gamma-glutamyl transferase (GGT), 5'nucleotidase (5' NT), total and conjugated bilirubin, albumin, INR, and ALP fractionated (hepatic).
Change from baseline in lipid parameters | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  Lipid parameters as measured by total cholesterol (TC), low-density lipoprotein cholesterol ( LDL-C), high-density lipoprotein cholesterol (HDL-C), calculated very low-density lipoprotein cholesterol (VLDL-C) and triglycerides (TG).
Change from baseline in liver stiffness measurement (LSM) | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  Assessed by vibration-controlled transient elastography (VCTE) using Fibroscan®
Change from baseline in pruritus | At Week 26, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  Based on PBC Worst Itch Numeric Rating Scale (NRS) score in participants with baseline PBC Worst Itch NRS score ≥4.
Proportion of responders in PBC Worst Itch NRS according to clinically meaningful change from baseline | At Week 26 and at Week 52 and every 26 weeks until the end of study (up to 6 years)
  At least 30% reduction; and one point, two points or three points decrease in score in participants with a baseline NRS score ≥4.
Proportion of participants with no worsening of pruritus from baseline | At Week 26 and at Week 52 and every 26 weeks until the end of study (up to 6 years)
Change from baseline in 5D-Itch scale | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  Questionnaire that assesses symptoms in terms of 5 domains: degree, duration, direction, disability and distribution. Participants rate their symptoms over the preceding 2-week period on a 1 to 5 scale, with 5 being the most affected.
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 7a scores | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  PROMIS Fatigue Short Form 7a scores consists of 7 items that measure both the experience of fatigue and the interference of fatigue on daily activities over the past week. Response options are on a 5-point Likert scale, ranging from 1 to 5. Scores can range from 7 to 35, with higher scores indicating greater fatigue.
Change from baseline in Epworth Sleepiness Scale (ESS). | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  Self-administered questionnaire that consists of 8 questions asking to rate how likely it is to fall asleep in different situations commonly encountered in daily life (each question can be scored from 0 to 3 points; '0' indicates no sleepiness, '3' indicates significant sleepiness). It provides a total score which has been shown to relate to the participant's level of daytime sleepiness (total score range 0-24 points).
Change from baseline in PBC-40. | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  40-item questionnaire that assesses symptoms across 6 domains: fatigue, emotional and social, cognitive function, general symptoms and itch. Participants respond on a verbal response scale, depending on the section options range from 'never' / 'not at all' / 'strongly disagree' to 'always' / 'very much' / 'strongly agree'. Six items (3/3 in the itch domain, 2/10 in the social domain, and 1/7 in the general symptoms domain) also include a 'does not apply' option. A score for each domain is provided (but a total score is not calculated), with each verbal response scale correlating to a score of 1 to 5 per item (0 to 5 on items with a 'does not apply' option) with 5 being the most affected (greatest burden).
Change from baseline in EuroQol 5-dimensional 5-level questionnaire (EQ-5D-5L) | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  Self-administered standardised questionnaire that assesses the 5-dimensions of mobility, self-care, usual activities, pain/discomfort, anxiety/depression descriptively (each dimension has 5 levels) and the overall health state via an EQ Visual Analogue Scale (VAS).
Change from baseline in Patient Global Impression of Severity (PGI-S) | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
  A 1-item, 5-point scale designed to assess the participant's impression of change in disease severity since the baseline visit
Patient Global Impression of Change (PGI-C) | At Week 4, Week 13, Week 26, Week 39, and Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)]
  A 1-item, 5-point scale designed to assess the participant's impression of change in disease severity since the baseline visit
Time to the first occurrence of each of individual adjudicated clinical outcome events | At Week 4, Week 13, Week 26, Week 39, Week 52, Week 78 and every 26 weeks until the end of study (up to 6 years)
Percentage of participants who experience Treatment Emergent Adverse Events (TEAEs), treatment related TEAEs, Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs). | From baseline to end of study (up to 6 years)
  An Adverse Event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AESIs are AEs that may not be serious but are of special importance to a particular drug or class of drugs.
Percentage of participants who develop clinically significant changes from baseline in physical examination findings | From baseline to end of study (up to 6 years)
  Clinically significant change in physical examination findings will be reported. The clinical significance will be graded by the investigator.
Percentage of participants who develop clinically significant changes from baseline in vital signs | From baseline to end of study (up to 6 years)
  Clinically significant change in vital signs will be reported. The clinical significance will be graded by the investigator.
Percentage of participants with clinically significant changes in laboratory parameters (blood chemistry, hematology, liver tests, renal tests (including urinalysis). | From baseline to end of study (up to 6 years)
  Clinically significant change in laboratory parameters will be reported. The clinical significance will be graded by the investigator.
Percentage of participants who develop clinically significant changes from baseline in ECG readings | From baseline to end of study (up to 6 years)
  Clinically significant change in ECG readings. The clinical significance will be graded by the investigator.
Change from baseline in fasting plasma glucose (FPG) Levels | At Week 52 and every 26 weeks until the end of study (up to 6 years)
Change from baseline in serum markers of bone turnover and in bone mineral density (hip and lumbar) | At Week 52 and every 26 weeks until the end of study (up to 6 years)
  Assessed by dual-energy X-ray absorptiometry (DEXA) scanning.
Area under the plasma concentration-time curve from time 0 to 24 hours: AUC0-24 | At Week 4
Maximum (peak) plasma drug concentration: Cmax | At Week 4
Time to reach maximum (peak) plasma concentration following drug administration): Tmax | At Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical, Director, Study Director — Ipsen
Locations (16):
- Japan (16):
  - Nippon Medical School - Chiba Hokusoh Hospital, Chiba
  - Fukushima Medical University Hospital, Fukushima
  - Chugoku Rosai Hospital, Hiroshima
  - Teine Keijinkai Hospital, Hokkaido
  - Kagawa University Hospital, Kagawa
  - Kagoshima University Hospital, Kagoshima
  - Shinshu University Hospital, Nagano
  - National Hospital Organization Nagasaki Medical Center, Nagasaki
  - Nara Medical University Hospital, Nara
  - Nagaoka Red Cross Hospital, Niigata
  - Niigata University Medical & Dental Hospital, Niigata
  - National Hospital Organization Osaka National Hospital, Osaka
  - Hamamatsu University Hospital, Shizuoka
  - Juntendo University Hospital, Tokyo
  - Teikyo University Hospital, Tokyo
  - Tokyo Metropolitan Komagome Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/